CLINICAL TRIAL: NCT07324356
Title: The Effect of Face-to-Face and Group Education Given to Mothers on Their Attitudes and Decisions Regarding Childhood Vaccinations
Brief Title: Effects of Individual and Group Education on Mothers' Attitudes and Decisions About Childhood Vaccination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Songül Çolak, Midwifery, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Istanbul University-Cerrahpa
Record Dates: First submitted 2025-11-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Childhood Immunization
Keywords: Vaccine hesitancy, Vaccination attitude, Vaccine education
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: This study will be carried out as a randomized controlled experimental study to determine the effect of face-to-face and group education given to mothers regarding childhood vaccinations on their attitudes and decisions about vaccination. Mothers who have children within the age range in which childhood vaccinations are administered will be contacted and informed about the purpose and scope of the study, and they will be asked whether they agree to participate. Mothers who consent to participate will be randomly assigned into three groups using computer-assisted randomization (https://www.random.org/
  ): Group 1: Mothers receiving individual face-to-face education, Group 2: Mothers receiving group education, and Group 3: Control group (receiving the routine unit-based information).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Mothers receiving individual face-to-face education (Experimental): After identifying eligible mothers, they will be contacted by phone and informed about the study. Mothers who agree to participate will be invited to the Family Health Center (FHC). Before the training, the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered.
  The first session of individual face-to-face education will be conducted using pre-prepared training content. An educational brochure related to the training content will be provided. After the session, the same forms and scales will be re-administered.
  Two weeks later, a second individual training session will be conducted to review and reinforce the previous education, and mothers' questions will be answered. Following the session, the data collection form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered again.
  Interventions: Behavioral: Vaccination attitude
- Group 2: Mothers receiving group education (Experimental): After identifying eligible mothers, they will be contacted by phone and informed about the study. Mothers who agree to participate will be invited to the Family Health Center (FHC) on scheduled dates for group training sessions. Before the training, the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered.
  The first group education session will be conducted using pre-prepared training content, and an educational brochure will be provided. After the session, the same forms and scales will be re-administered.
  Two weeks later, a second group education session will be conducted to review and reinforce the previous education, and participants' questions will be answered. After the session, the data collection form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered again.
  Interventions: Behavioral: Vaccination attitude
- Group 3: Control group (receiving the routine unit-based information) (No Intervention): After identifying mothers who will receive routine informational training at the Family Health Center (FHC), they will be contacted by phone and informed about the study. Mothers who agree to participate will be invited to the FHC. Before the routine training, the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered.
  Routine training provided by the FHC will then be conducted. After the training, the same data collection form and scales will be re-administered.
  Two weeks later, participants will be invited again to receive routine training once more, and following the training, the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered again.

INTERVENTIONS:
Behavioral: Vaccination attitude — This study was planned to determine the effect of face-to-face and group education given to mothers regarding childhood vaccinations on their attitudes and decisions about vaccination. It is thought that the education provided will help eliminate mothers' misconceptions and false beliefs about vaccines in the short term and contribute to positive changes in their attitudes and decisions regarding vaccination. Moreover, it is anticipated that, in the long term, this intervention will contribute to achieving better immunization rates and protecting children from vaccine-preventable diseases. This study is also important in terms of emphasizing the midwife's role in protecting and improving infant and community health.
  Arms: Group 1: Mothers receiving individual face-to-face education; Group 2: Mothers receiving group education

SUMMARY:
This study was planned to determine the effect of face-to-face and group education given to mothers regarding childhood vaccinations on their vaccination attitudes and decisions. It is believed that the education provided will help eliminate mothers' misconceptions and false beliefs about vaccines in the short term, and contribute to positive changes in their attitudes and decisions regarding vaccination. Moreover, it is anticipated that in the long term, this intervention will contribute to achieving better immunization rates and protecting children from vaccine-preventable diseases. This study is also important in terms of emphasizing the role of midwives in protecting and improving infant and community health.This study will be carried out as a randomized controlled experimental study to determine the effect of face-to-face and group education given to mothers regarding childhood vaccinations on their attitudes and decisions about vaccination. Mothers who have children within the age range in which childhood vaccinations are administered will be contacted and informed about the purpose and scope of the study, and they will be asked whether they agree to participate. Mothers who consent to participate will be randomly assigned into three groups using computer-assisted randomization (https://www.random.org/

): Group 1: Mothers receiving individual face-to-face education, Group 2: Mothers receiving group education, and Group 3: Control group (receiving the routine unit-based information).

DETAILED DESCRIPTION:
Experimental Group 1

(Group 1: Mothers Receiving Individual Face-to-Face Education)

After identifying the mothers to whom the education will be provided, they will be contacted by phone using their contact information and informed about the study. Mothers who agree to participate will be invited to the Family Health Center (FHC). Before the education, the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered.

The first session of individual face-to-face education will then be conducted using previously prepared educational content. An educational brochure related to the content of the training will be given to the mothers. After the education session, the data collection form, vaccine attitudes scale, and vaccine hesitancy scale will be administered again.

The second education session will be conducted two weeks later. In this session, the previously provided information will be reviewed and reinforced, and the mothers' questions will be answered. Following the session, the data collection form, vaccine attitudes scale, and vaccine hesitancy scale will be re-administered.

Experimental Group 2

(Group 2: Mothers Receiving Group Education)

After identifying the mothers to whom the education will be provided, they will be contacted by phone and informed about the study. Mothers who agree to participate will be invited to the FHC to attend group education sessions scheduled at appropriate dates and times. Before the education, the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered.

The first session of the group education will be conducted using previously prepared educational content. An educational brochure related to the content of the training will be given to the mothers. After the education session, the data collection form, vaccine attitudes scale, and vaccine hesitancy scale will be administered again.

The second education session will be conducted two weeks later. In this session, the previously provided information will be reviewed and reinforced, and the mothers' questions will be answered. Following the session, the data collection form, vaccine attitudes scale, and vaccine hesitancy scale will be re-administered.

Control Group

(Group 3: Mothers Receiving Routine Education)

After identifying the mothers who will receive routine education at the FHC, they will be contacted by phone and informed about the study. The mothers will be invited to the FHC, where the Data Collection Form, Vaccine Attitudes Scale, and Vaccine Hesitancy Scale will be administered prior to the education.

Subsequently, the routine education provided by the FHC will be delivered, and an educational brochure will also be given to the mothers in the control group. After the education, the data collection form, vaccine attitudes scale, and vaccine hesitancy scale will be administered again.

Two weeks later, the mothers will be invited to the FHC again, the routine education will be repeated, and after the education, the data collection form, vaccine attitudes scale, and vaccine hesitancy scale will be re-administered.

ELIGIBILITY:
Inclusion Criteria:

* Being registered at Rumeli Family Health Center, Bağcılar, Istanbul
* Ability to speak and understand Turkish
* Ability to read and write
* Having a child within the age range covered by the national vaccination schedule (0-13 years)
* Being 18 years of age or older
* Willingness to participate in the study

Exclusion Criteria:

* Not attending one or more of the educational sessions

Participating in any training other than the vaccination education program

Failing to complete the data collection forms in full

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 75 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Vaccine Opposition Scale | 6 month
  The total score of the long form ranges from 21 to 105, while the total score of the short form ranges from 12 to 60. Higher scores on the scale indicate higher levels of vaccine hesitancy among participants."The long form of the scale demonstrated high internal consistency (Cronbach's alpha = 0.905)."
Vaccine Attitudes Scale | 6 month
  Each item on the Vaccine Attitudes Scale is scored as agree = 1, undecided = 2, and disagree = 3. The total score is calculated by summing the item scores. The possible total score ranges from 11 to 33, where a score of 11 indicates a positive parental attitude toward vaccination, and a score of 33 indicates a negative attitude toward vaccination.
  The scale does not have a cut-off point. As the total score increases, parental vaccine hesitancy increases, reflecting a more negative attitude toward vaccination.
  "The Turkish version of the scale demonstrated acceptable internal consistency (Cronbach's alpha = 0.66)."
Data Collection Form | 6 month
  This form was developed by the researcher and the advisor based on the relevant literature (Yorulmaz et al., 2024; Ünsal, 2020; Yiğit et al., 2020; Hazır, 2018) and consists of 27 questions. It will be used in the study to determine mothers' demographic and descriptive characteristics and their decisions regarding vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Songül ÇOLAK, Principal Investigator — Istanbul Provincial Directorate of Health
Locations (1):
- Rumeli Aile Sağlığı Merkezi, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No